CLINICAL TRIAL: NCT03280095
Title: A Randomised, Open-label, Three-treatment, Single Dose, Crossover Study Investigating the Bioequivalence of Co-codamol 15/500mg Capsules With a Co-codamol 30/500mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Co-codamol 15mg/500mg Capsules vs Co-codamol 30mg/500mg Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galen Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BKE12814; 2014-003334-12 (EudraCT Number)
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — acetaminophen, codeine drug combination; Tablets

ARMS (3):
- Treatment 1 (Experimental): One capsule of test product (co-codamol 15mg/500mg capsule) containing 15mg codeine phosphate hemihydrate and 500mg paracetamol.
  Interventions: Drug: co-codamol 15mg/500mg capsule
- Treatment 2 (Experimental): Two capsules of test product (co-codamol 15mg/500mg capsule), each containing 15mg codeine phosphate hemihydrate and 500mg paracetamol (i.e. a total dose of 30mg codeine phosphate hemihydrate and 1000mg paracetamol).
  Interventions: Drug: co-codamol 15mg/500mg capsule
- Treatment 3 (Active Comparator): One tablet of reference product (co-codamol 30mg/500mg tablet) containing 30mg codeine phosphate hemihydrate and 500mg paracetamol.
  Interventions: Drug: co-codamol 30mg/500mg tablet

INTERVENTIONS:
Drug: co-codamol 15mg/500mg capsule
  Arms: Treatment 1; Treatment 2
Drug: co-codamol 30mg/500mg tablet
  Arms: Treatment 3

SUMMARY:
The purpose of this study is to compare the bioavailability of co-codamol 15mg/500mg capsules (test product) and co-codamol 30mg/500mg tablets (reference product).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18-45 (both inclusive), as determined by medical history, physical examination, laboratory test values, vital signs and 12-lead ECGs at screening.
* Non-smokers from at least three months before receiving the first dose of study drug and for the duration of the study.
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Able to voluntarily provide written informed consent to participate in the study.
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol, as confirmed during the informed consent process.
* Female volunteers of child-bearing potential and less than one year postmenopausal must have a negative serum pregnancy test and be non-lactating.
* Female volunteers who have been post-menopausal for more than one year and have elevated serum follicle stimulating hormone (FSH) or are treated with hormone replacement therapy (HRT) or female volunteers who have been permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy).
* Male volunteers and female volunteers of child-bearing potential who are sexually active must use two highly effective methods of contraception with their partners throughout the study and for 30 days after completion of the study (female volunteers) or 90 days after completion of the study (male volunteers). Acceptable methods include: condom or occlusive cap (diaphragm or cervical/ vault caps) with spermicidal foam/ gel/ film/ cream/ suppository; male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); established use of oral, injected or implanted hormonal methods of contraception and placement of an intrauterine device or intrauterine system. True abstinence is an acceptable method only where this is already established as the volunteer's preferred and usual lifestyle.
* Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
* The volunteer's primary care physician has confirmed within the last 12 months that there is nothing in their medical history that would preclude their enrolment into a clinical study.
* Volunteers should be cautioned that codeine may impair mental and/or physical abilities, therefore it may affect their ability to drive or operate machinery for up to approximately 24 hours post-dose.

Exclusion Criteria:

* Volunteers with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, urogenital (including benign prostatic hypertrophy), haematological, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or current infection.
* Laboratory values at screening which are deemed to be clinically significant, unless agreed in advance by the Sponsor's Medical Representative and Principal Investigator.
* Female volunteers who are pregnant or lactating.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Current or history of drug or alcohol abuse or a positive drugs of abuse or alcohol test at screening or check-in.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Any clinically significant illness within 30 days prior to study drug administration.
* Donation of blood or blood products within 90 days prior to study drug administration, or at any time during the study, except as required by this protocol.
* Volunteers who have a history or presence of any significant drug allergy, including a history of hypersensitivity to paracetamol, codeine phosphate hemihydrate, any related drugs, or any of the excipients contained in the formulations.
* Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 14 days prior to study drug administration until the end of the study, with the exception of Investigator approved contraceptives and HRT.
* Volunteers with inadequate venous access to allow collection of blood samples as required by this protocol.
* Strenuous exercise, as judged by the Investigator, within 72 hours prior to screening, within 72 hours prior to study drug administration and for the duration of the study until after the post-study medical.
* Weekly alcohol intake exceeding the equivalent of 14 units per week for females or 21 units per week for males.
* Consumption of alcoholic beverages within 48 hours prior to study drug administration and during study confinement.
* Consumption of caffeine or xanthine-containing products within 24 hours prior to study drug administration and during study confinement.
* Consumption of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade or other products containing grapefruit or Seville oranges within 7 days prior to study drug administration, during study confinement and during the wash-out periods.
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2014-12-12 (Actual); Study Completion 2014-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum measurable plasma concentration (Cmax) | 0 to 36 hours post-dose
  Cmax and AUC0-t will be used to calculate bioequivalence of the test product (Treatment 1) vs reference product (Treatment 3) for paracetamol, and test product (Treatment 2) vs reference product (Treatment 3) for codeine.
Area under the plasma concentration versus time curve from drug administration to last observed concentration at time t (AUC0-t) | 0 to 36 hours post-dose
  Cmax and AUC0-t will be used to calculate bioequivalence of the test product (Treatment 1) vs reference product (Treatment 3) for paracetamol, and test product (Treatment 2) vs reference product (Treatment 3) for codeine.

SECONDARY OUTCOMES:
Adverse events, including laboratory parameters. | 23 days
  The safety of volunteers will be monitored by recording adverse events, including laboratory parameters.
Time of maximum measured plasma concentration (Tmax) | 0 to 36 hours post-dose
  The pharmacokinetic parameter Tmax will be measured for test and reference products.
Elimination rate constant (Kel) | 0 to 36 hours post-dose
  The pharmacokinetic parameter Kel will be measured for test and reference products.
Elimination or terminal half-life (t1/2) | 0 to 36 hours post-dose
  The pharmacokinetic parameter t1/2 will be measured for test and reference products.
Area under the plasma concentration versus time curve from time zero extrapolated to infinity (AUC0-∞) | 0 to 36 hours post-dose
  The pharmacokinetic parameter AUC0-∞ will be measured for test and reference products.

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, MD, Principal Investigator — BioKinetic Europe Ltd
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom